CLINICAL TRIAL: NCT01297205
Title: Open Label, Single-Center, Phase 1 Clinical Study to Evaluate the Safety and the Efficacy of PNEUMOSTEM® Treatment in Premature Infants With Bronchopulmonary Dysplasia
Brief Title: Safety and Efficacy Evaluation of PNEUMOSTEM® Treatment in Premature Infants With Bronchopulmonary Dysplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-CR-006
Record Dates: First submitted 2011-02-11; First posted 2011-02-16 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Human Umbilical Cord Blood Derived Mesenchymal Stem Cells; Bronchopulmonary dysplasia; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PNEUMOSTEM® (Experimental)
  Interventions: Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells — Dose A - 10 million cells per kg Dose B - 20 million cells per kg Single intratracheal administration
  Other Names: PNEUMOSTEM®

SUMMARY:
PNEUMOSTEM® is human umbilical cord blood derived mesenchymal stem cells and it is intended to treat premature infants with bronchopulmonary dysplasia. This study is to assess the safety and the efficacy of this study drug.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is most common cause of death of children who were born prematurely, with low birth weights. In addition, many children who were recovered from this disease are suffering from many side effects such as prolonged hospitalization, pulmonary hypertension, and failure to thrive.

The purpose of BPD treatment is to make a baby be able to do spontaneous breathing and to spontaneous breathing a baby needs much energy and because of this a baby may have difficulty to feed. For this reason, medication with steroid, diuretic and respiratory drugs are currently used. However, there is no effective cure so far.

It has been reported that bone marrow derived mesenchymal stem cells (BM-MSC) can differentiate to pulmonary epithelial and pulmonary endothelial cells. Some animal studies showed that BM-MSC differentiated to bronchial cells and type 2 pneumocytes in rats with pneumonia and improve the fibrosis that occur after administration of bleomycin. Based on the findings, it is considered that mesenchymal stem cell therapy can help regenerate the damaged lung as well as BPD that cause lung inflammation, fibrosis, deficiency of type 2 pneumocytes, and so on.

PNEUMOSTEM® is human umbilical cord blood derived mesenchymal stem cells and it is intended to treat premature infants with BPD. The main purpose of this study is to evaluate the safety and the tolerability of this study drug and to establish the maximum toxicity dose. The latent efficacy will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight range: 500g~1250g
* Fetal gestational age: 23 weeks to 29 weeks
* Premature infants who cannot do spontaneous breathing, which ventilation rate is less than 12 breaths per min of ventilation rate and 25% of oxygen demand
* Premature infants who does not improve the breathing or worse within 24 hours prior to enrollment of this study
* Written consent form signed by a legal representative or a parent

Exclusion Criteria:

* Cyanotic or acyanotic congenital heart diseases except patent ductus arteriosus
* Severe lung malformation (i.e. Pulmonary hypoplasia, congenital diaphragmatic hernia, congenital cystic lung disease)
* Severe lung malformation with chromosome anomalies (i.e. Edward syndrome, Patau syndrome, Down syndrome, etc) or severe congenital malformation (Hydrocephalus, Encephalocele, etc)
* Severe congenital infection (i.e. Herpes, Toxoplasmosis, Rubella, Syphilis, AIDS, etc)
* CRP > 30 mg/dL; Severe sepsis or shock
* Premature infants who is going to or expected to have surgery 72 hours before/after this study drug administration
* Surfactant administration within 24 hours prior to this study drug administration
* Severe intracranial hemorrhage ≥ grade 3 or 4
* Premature infants who have active pulmonary hemorrhage or active air leak syndrome at the time point of screening
* History of other clinical studies as a participant
* Premature infants who are allergic to Gentamicin
* Premature infants who is considered inappropriate by the investigators

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participant with adverse reaction | 12 weeks from the day of treatment
  Number of paitents with normal rage of vital signs and laboratory examination Chest x-ray result, Duration of ventilator dependence, Duration of CPAP treatment, Duration of intubation, Occurrence of pneumothorax, Occurrence of intraventricular hemorrhage, Postnatal steroid use (%), Dose of surfactant (%) Cumulative duration of oxygen use

SECONDARY OUTCOMES:
Incidence of BPD at 36 Week's postmenstrual age | 36 week's postmenstrual age
  Incidence of BPD at 36 Week's postmenstrual age (PMA)and 28 week's PMA Survival rate at 28 days after birth and 36 week's PMA

CONTACTS AND LOCATIONS:
Overall Officials: Won-Soon Park, M.D., PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chang YS, Ahn SY, Yoo HS, Sung SI, Choi SJ, Oh WI, Park WS. Mesenchymal stem cells for bronchopulmonary dysplasia: phase 1 dose-escalation clinical trial. J Pediatr. 2014 May;164(5):966-972.e6. doi: 10.1016/j.jpeds.2013.12.011. Epub 2014 Feb 6. PMID 24508444